CLINICAL TRIAL: NCT06469021
Title: Effectiveness of Rehabilitation with Technology-Based Systems in Adolescent Idiopathic Scoliosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: hande tunc (Other)
Responsible Party: Sponsor-Investigator, hande tunc, Doctor of Philosophy Candidate (PhD(c)), Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-3224
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Scoliosis; Adolescence
Keywords: Scoliosis; Virtual Reality; Technology Based Rehabilitation
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group: (Active Comparator): The control group will perform the structured three-dimensional scoliosis exercise, core stabilization, and balance exercise with conventional methods at the clinic and home setting for twenty-four weeks. In the clinical setting, patients will perform their exercise for 2 days a week for 12 weeks, 1 day a week for the next 12 weeks, under the supervision of a physiotherapist. Patients will be asked to perform their exercises as a home exercise program on the remaining days (home exercise program 3 days a week for the first 12 weeks, 4 days a week after week 12).
  Interventions: Other: Conservative Approach
- Rehabilitative Game Based Exercise Group (Experimental): The Rehabilitative Game-Based Exercise group will perform the structured three-dimensional scoliosis exercise with conventional methods similar to the control group. Differently, technology-based systems (BeCure Systems) will be used in the implementation of core stabilization and balance exercises. Patients will be asked to perform their exercises as a home exercise program on the remaining days (home exercise program 3 days a week for the first 12 weeks, 4 days a week after week 12).
  Interventions: Other: Rehabilitative Game Therapy

INTERVENTIONS:
Other: Conservative Approach — Structured scoliosis exercises will be prescribed by the physiotherapist according to the severity of the curvature and cosmetics of the individuals. In a one session period, 5-minute warm-up and cool-down periods, 20 minutes of scoliosis exercises, 10 minutes of core stabilization exercises and 10 minutes of balance training will be applied. The exercises will start from an easy level and the level of difficulty will be gradually increased. The assessments will be evaluated in three stages: at the beginning of treatment, at the third month of treatment and at the end of treatment (sixth month).
  Arms: Control Group:
Other: Rehabilitative Game Therapy — Structured scoliosis exercises will be prescribed by the physiotherapist according to the severity of the curvature and cosmetics of the patients and will be applied to the patients with a conventional approach. In a one-session period, 5-minute warm-up and cool-down periods, 20 minutes of scoliosis exercises, 10 minutes of core stabilization exercises, and 10 minutes of balance training will be applied in the clinical setting. Home exercises will be performing with the SmartPose system differently from the control group. The SmartPose system is a special software system that enables the user to perform movements with a tablet or phone without the need for any sensors.
  Arms: Rehabilitative Game Based Exercise Group

SUMMARY:
The aim of this study was to investigate the effect of technology-based exercises on treatment success in adolescents with idiopathic scoliosis.

Within the scope of the study, thirty patients with AIS will be randomly allocated to two groups. The control group will apply a program with conventional approaches consisting of a combination of structured three-dimensional scoliosis exercises, core stabilization and balance exercises. Patients in the intervention group will perform structured three-dimensional scoliosis exercises, core stabilization and balance exercises similarly to the control group. However, patients in the intervention group will perform core stabilization and balance exercises with virtual reality games for twenty-four weeks. Patients' Cobb angle, Pediatric Berg Balance Scale (balance), Posterior Trunk Asymmetry Index (POTSI) (cosmetic), Walter Reed Visual Assessment Scale (WRVAS)(cosmetic), System Usability Scale (system usability) and Physical Activity Participation Motivation Scale (PAPMS) (motivation) parameters will be assess at the beginning of treatment, third and six month.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional structural deformity in growing children, not associated with a cause, in which lateral deviation of the spine over 10° is accompanied by rotation. The magnitude of the Cobb angle is used to classify the severity of scoliosis. In immature AIS cases, if the Cobb angle is between 25°-40°, bracing and exercise therapy is applied. Exercise in AIS is performed to reduce clinical symptoms, improve cosmetics and prevent curve progression. Corrective exercises based on sensorimotor and kinesthetic principles include self-correction in front of a mirror, three-dimensional breathing techniques and home exercise programs.

Virtual reality applications (VRA) are three-dimensional computer simulations that give the individual the feeling of "being anywhere" and provide various information (light, sound and others) to the sensory organs. VRS is based on motor learning principles. The possibility of repetitive movements and computer feedback results in positive changes at the cortical level. In addition, the virtual environment increases the motivation of the individual and ensures active participation in the treatment.

A review of the literature reveals that there are very limited studies on technology-based applications or virtual reality in scoliosis rehabilitation. To the best of our knowledge, it has been observed that there is no long-term rehabilitation protocol applied on the basis of rehabilitative game therapy in AIS rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Adolescent Idiopathic Scoliosis,
* Girls and boys aged between 10-15,
* Being the Cobb angle between 25-40 degrees,
* Being using three dimensional brace,
* Being immature (Risser 0-2 or Sanders 1-4 phase)
* Regular follow-ups (0-3-6 months)

Exclusion Criteria:

* Presence of previous spinal surgery,
* Progression resulting in the necessity of surgery,
* Participation in any exercise therapy program,
* Playing sports at a professional level,
* Cardiac and respiratory dysfunction and/or concomitant systemic disease,
* Health (mental, orthopedic) problems that prevent exercise

Ages: 10 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cobb Angle | At the beginning of the study and sixth month of the study
  In the treatment of scoliosis, the Cobb angle is considered the most important outcome for the evaluation of treatment efficacy. The Cobb angle is measured from anteroposterior graphs taken during standing. Measurements will be taken by a blinded assessor via SurgiMap web application to eliminate individual errors. Measurements will be made from radiographs taken at the beginning and sixth month of treatment because of the radiation exposure.
Posterior Trunk Symmetry Index (POTSI) | At the beginning of the study, third month and sixth month of the study
  POTSI is a method that makes it possible to evaluate the trunk asymmetry of an individual with AIS from the posterior and objectively scores the cosmetic effect. It is based on certain calculations performed on a posterior photograph of the individual. The score calculated in POTSI analysis consists of the sum of 6 indices. In order to prevent possible calculation errors and standardize the measurements, the cases will be evaluated with a mobile application named POTSIApp.
Walter Reed Visuel Assessment Scale (WRVAS) | At the beginning of the study, third month and sixth month of the study
  WRVAS is a scale that scores the severity of curvature by focusing on the person's perception of posture. It is divided into 7 parameters including body curvature, rib prominence, lumbar prominence, head-rib-pelvis positional relationship, head-pelvis relationship, shoulder level and scapula rotation. A high score means that the perceived deformity is high.

SECONDARY OUTCOMES:
Single Leg Balance Test | At the beginning of the study, third month and sixth month of the study
  One foot is lifted so that it does not touch the support leg, eyes are open at the beginning. The eyes are fixed in the direction of the head, the patient is asked to close his/her eyes and is expected to maintain his/her balance for 30 seconds. If the lifted leg touches the support leg, if the foot touches the floor, if there is bouncing or jumping, or if anything in the environment is touched for support, a balance disorder is considered.
The Physical Activity Participation Motivation Scale (PAPMS) | At the beginning of the study, third month and sixth month of the study
  The Physical Activity Participation Motivation Scale (PAPMS) is a Likert-type scale used to assess the motivation levels of individuals for physical activity. The scale consists of 3 sub-dimensions (individual reasons, environmental reasons and lack of reason dimension) and a total of 16 questions in 5-point Likert type. High values are associated with high motivation level.
The System Usability Scale (SUS) | At the beginning of the study, third month and sixth month of the study
  The System Usability Scale (SUS) is a scale used to evaluate usability. It is a 10-item Likert-type scale that can be used individually and allows general usability evaluation. High scores on the scale indicate that systems are usable.
Angle of Trunk Rotation | At the beginning of the study, third month and sixth month of the study
  The scoliometer is a specially designed inclinometer that is easy to use, inexpensive, reliable and practical for the clinical assessment of scoliosis. inexpensive, reliable and practical for the clinical assessment of scoliosis. Inside the scoliometer is a metal sphere that moves in the water bed and higher degrees indicates increased degree of body rotation. In the forward bending position, the scoliometer is placed vertically on the axial axis of the spine perpendicular to the spinous process of the vertebra and measured

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziosmanpasa Training and Reserach Hospital, Istanbul
  - Istanbul Medipol University, Istanbul

IPD SHARING:
Plan to Share IPD: No